CLINICAL TRIAL: NCT03710629
Title: A Prospective Observational Study to Explore Treatment Regimens and Clinical Outcomes of the NSCLC Patients With Different Driver Genes
Brief Title: A Study to Explore Treatment Regimens and Clinical Outcomes of the NSCLC Patients With Different Dirver Genes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GZH-Gene
Record Dates: First submitted 2018-07-10; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer, gene mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients with driver genes: NSCLC patients and driver genes
  Interventions: Other: Patients with driver genes

INTERVENTIONS:
Other: Patients with driver genes — Patients with driver genes

SUMMARY:
A single-center, non-interventional prospective observational study in the NSCLC patients with different driver genes

DETAILED DESCRIPTION:
The trial was designed as a single-center non-interventional prospective observational study to explore clinical treatments of the NSCLC patients with different driver genes, the impact factors of patient survivals, and the relevance of gene types, clinical treatments, and distribution of gene types. The follow-up visits, interactions between the investigators and patients, patient questionnaires/quality of life, and other patient information will be uploaded via mobile APP, and webchat every three months.

ELIGIBILITY:
Inclusion Criteria:

* The patients with lung cancer who were performed with next-generation sequencing (NGS) technology from 2015 to 2017;
* The patients who were at least 18 years;
* The pathologically diagnosed patients with non-small cell lung cancer (NSCLC)

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pathologically diagnosed patients with non-small cell lung cancer who were performed with NGS technology
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Differences in overall survival rates | 2018-2022
  Differences in overall survival rates of the NSCLC patients with various gene types

SECONDARY OUTCOMES:
Interaction impact between gene types and treatment modalities or regimens on disease-free survivals | 2018-2022
  Interaction impact between gene types and treatment modalities or regimens on disease-free survivals
Statuses of clinical treatment regimens | 2018-2022
  Statuses of clinical treatment regimens of the NSCLC patients
Relevance of gene types | 2018-2022
  Relevance of gene types and clinical characteristics of the NSCLC patients
Relevance of overall survival rates and gene types | 2018-2022
  Relevance of overall survival rates and gene types of the NSCLC patients
Impacts of disease-free survivals on gene types | 2018-2022
  Impacts of disease-free survivals on gene types of the NSCLC patients
Impacts of progression-free survivals | 2018-2022
  Impacts of progression-free survivals on gene types of the NSCLC patients
Impact factors of overall survivals | 2018-2022
  Impact factors of overall survivals of the NSCLC patients

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua Liang, Ph.D, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Wenhua of Liang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No